CLINICAL TRIAL: NCT01427738
Title: A Phase III, Open-Label, Randomized, Assessment-Blinded Clinical Trial to Compare the Safety and Efficacy of Gentian Violet Oral Solution to That of Nystatin Oral Suspension for the Treatment of Oropharyngeal Candidiasis in HIV-1 Infected Participants in Non-U.S. Settings
Brief Title: Gentian Violet Vs. Nystatin Oral Suspension for Treatment of Oropharyngeal Candidiasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5265; 1U01AI068636 (NIH); NCT01494129 (obsolete NCT alias)
Record Dates: First submitted 2010-11-03; First posted 2011-09-02 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Gentian Violet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Topical GV solution (Experimental): Topical GV 0.00165% solution (5 mL swish and gargle for 1 minute and expectorate [spit] 2 times per day [BID]) for 14 days
  Interventions: Drug: Gentian Violet
- Arm B: Nystatin oral suspension (Active Comparator): Nystatin oral suspension (5 mL of 100,000 units/mL swish for 1 minute and swallow 4 times per day [QID]) for 14 days
  Interventions: Drug: Nystatin oral suspension

INTERVENTIONS:
Drug: Gentian Violet — Participants were administered topical Gentian violet solution, orally, twice daily for 14 days.
  Arms: Arm A: Topical GV solution
Drug: Nystatin oral suspension — Participants were administered Nystatin oral suspension 4 times a day for 14 days.
  Arms: Arm B: Nystatin oral suspension

SUMMARY:
The purpose of this study was to see which one of two medicines (topical gentian violet [GV] or nystatin oral suspension) was better than the other in treating Oral Candidiasis (OC). This was measured by whether the study participant still had OC or sores in his/her mouth after 14 days of treatment. Also, safety and tolerability of GV and nystatin in the treatment of OC were assessed.

DETAILED DESCRIPTION:
A5265 was a phase III, open-label (both the researchers and participants know which treatment was being administered) clinical trial to compare the safety and efficacy of topical GV to that of oral nystatin suspension. Male and female HIV-1 positive participants ≥ 18 years of age were randomized (as if by the toss of a coin) with equal probability and stratified by CD4+ T-cell counts and the use of antiretroviral therapy at the time of study entry to receive either topical GV solution (5 mL swish and gargle for 1 minute and spit two times daily) or nystatin oral suspension (5 mL swish for 1 minute and swallow four times daily) for 14 days. Therapy was considered as failed if participants have no clinical improvement (assessed by severity of pseudomembranous candidiasis) during either treatment regimen. Evaluation of signs and symptoms of oral candidiasis was done by an evaluator who was blinded to the treatment assignment. A total of 494 participants was expected to enroll in the study but due to early study closure only 221 enrolled; and participants are expected to be on the study for about 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.
* Pseudomembranous candidiasis documented by a complete oral exam (i.e., white or yellow spots or plaques with an underlying erythematous base, located in any part of the oral cavity) at the screening visit. Participants with documented angular chelitis and/or erythematous candidiasis without pseudomembranous candidiasis were not eligible to enroll in the study.
* If on an antiretroviral therapy (ART), initiation of regimen at least 12 weeks prior to study entry, and willingness of participant to remain on current ART regimen until the study-defined 14-day treatment period was complete. NOTE: Participants who were not ART-naïve and not on ART were eligible to participate in the study if they did not intend to initiate ART during the study- defined 14-day treatment period.
* CD4+ cell count obtained within 30 days prior to study entry at a DAIDS-approved laboratory.

Exclusion Criteria:

* Documented or presumptive signs or symptoms of esophageal candidiasis (e.g., dysphagia) during the screening period unless endoscopic examination of the esophagus was performed, and fungal esophagitis were excluded.
* Use of any investigational drug currently or within 30 days prior to study entry. NOTE: For purposes of this study, drugs available under an FDA-authorized expanded access program was NOT considered investigational.
* Concurrent vaginal candidiasis within 21 days prior to study entry.
* Use of inhaled or systemic corticosteroids within 14 days prior to study entry.
* Use of any antifungal agents within 30 days prior to study entry.
* Anticipated need for systemic or oral/topical antifungal agents for other diagnoses within the study-defined 14-day treatment period.
* Intend to initiate ART during the screening period, at study entry, or within the study-defined 14-day treatment period.
* Intend to use any additional oral topical treatments within the study- defined 14-day treatment period.
* Known allergy/sensitivity or any hypersensitivity to components of study drugs or their formulation.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serious illness, in the opinion of the site investigator, requiring systemic treatment.
* Hospitalization within 30 days prior to study entry for HIV or HIV-related conditions.
* Previous or current history of porphyria.
* Presence of oral warts during the screening period or at the study entry visit before randomization.
* Current wearing of full dentures or a maxillary partial denture at study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Salata, MD, Study Chair — Case CRS; James G Hakim, MD, Principal Investigator — UZ- Parirenyatwa CRS; Tim Hodgson, MD, Principal Investigator — Eastman Dental Hospital; Richard J Jurevic, DDS, PhD, Principal Investigator — Case CRS; Pranab K Mukherjee, PhD, MSc, Principal Investigator — Case CRS; Cissy M Kityo, MBChB, MSc, Principal Investigator — JCRC CRS; Rana Traboulsi, MD, Principal Investigator — Case CRS; Srikanth P Tripathy, MD, MBBS, Principal Investigator — NARI Pune CRS; Mahmoud A Ghannoum, Phd, MSc, Principal Investigator — Case Western Reserve University
Locations (10):
- Botswana (2):
  - Gaborone Prevention/Treatment Trials CRS (12701), Gaborone
  - Molepolole Prevention/Treatment Trials CRS (12702), Molepolole
- India (2):
  - BJ Medical College CRS (31441), Pune, Maharashtra
  - National AIDS Research Institute Pune CRS (11601), Pune, Maharashtra
- Kenya (2):
  - AMPATH at Moi Univ. Teaching Hosp. Eldoret CRS (12601), Eldoret
  - Walter Reed Project - Kenya Med. Research Institute Kericho CRS (12501), Kericho
- College of Med. JHU CRS (30301), Blantyre, Malawi
- Durban Adult HIV CRS (11201), Durban, South Africa
- Joint Clinical Research Centre (JCRC) (12401), Kampala, Uganda
- UZ-Parirenyatwa CRS (30313), Harare, Zimbabwe

REFERENCES:
- [Derived] Mukherjee PK, Chen H, Patton LL, Evans S, Lee A, Kumwenda J, Hakim J, Masheto G, Sawe F, Pho MT, Freedberg KA, Shiboski CH, Ghannoum MA, Salata RA; Oral HIVAIDS Research Alliance (OHARA)AIDS Clinical Trials Group (ACTG) 5265 Team. Topical gentian violet compared with nystatin oral suspension for the treatment of oropharyngeal candidiasis in HIV-1-infected participants. AIDS. 2017 Jan 2;31(1):81-88. doi: 10.1097/QAD.0000000000001286. PMID 27677161

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Topical GV Solution: Topical GV 0.00165% solution (5 mL swish and gargle for 1 minute and expectorate [spit] 2 times per day [BID]) for 14 days
  Gentian Violet: Participants will be administered topical Gentian violet solution, orally, twice daily for 14 days.
- Arm B: Nystatin Oral Suspension: Nystatin oral suspension (5 mL of 100,000 units/mL swish for 1 minute and swallow 4 times per day [QID]) for 14 days
  Nystatin oral suspension: Participants will be administered Nystatin oral suspension 4 times a day for 14 days.
Period: Overall Study
Arm/Group | Arm A: Topical GV Solution | Arm B: Nystatin Oral Suspension
Started | 110 | 111
Completed | 91 | 90
Not Completed | 19 | 21
Not completed — Death | 12 | 9
Not completed — Severe debilitation, unable to continue | 0 | 1
Not completed — Subject unable to get to clinic | 5 | 2
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Subject not willing to adhere to reqs | 1 | 2
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Population: All participants who enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Topical GV Solution | Arm B: Nystatin Oral Suspension | Total
Number analyzed (Participants) | 110 | 111 | 221
Age, Customized [Number; unit: participants]
  10-19 years | 0 | 1 | 1
  20-29 years | 17 | 30 | 47
  30-39 years | 54 | 52 | 106
  40-49 years | 21 | 17 | 38
  50-59 years | 16 | 9 | 25
  Over 60 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 66 | 128
  Male | 48 | 45 | 93
Race/Ethnicity, Customized [Number; unit: participants]
  Black Non-Hispanic | 97 | 106 | 203
  Asian, Pacific Islander | 13 | 5 | 18
Antiretroviral Therapy Usage [Number; unit: participants]
  On ART | 27 | 28 | 55
  Not on ART | 83 | 83 | 166
CD4 Count [Number; unit: participants]
  0-200 cells/microliter | 87 | 88 | 175
  > 200 cells/microliter | 23 | 23 | 46
HIV RNA Viral Load [Mean (Standard Deviation); unit: log10(copies/ml)] | 4.89 (1.31) | 5.03 (1.21) | 4.96 (1.26)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Efficacy
Description: The primary endpoint is clinical efficacy defined as cure (absence of lesions) or improvement (a decrease in severity of lesions) after 14 days of treatment. The oral cavity will be split arbitrarily into 6 sites: left lower and upper labial mucosa and buccal mucosa, right lower and upper labial mucosa and buccal mucosa, hard palate, soft palate, tongue (dorsum, lateral, and ventral), and floor of mouth. Severity is scored using a scoring system from 0 to 3 (0 corresponds to absence of lesions, and 3 corresponds to presence of extensive confluent lesions) which leads to a composite severity score ranging from 0 to 18 after adding up the scores from all 6 sites. Complete success is assigned if the composite score after treatment equals to 0. Improved/partial response is assigned if the composite score after treatment is less than the baseline score. The blinded evaluator scores the severity of lesions by examining different lesion characteristics.
Time Frame: After 14 days of treatment
Population: Out of 221 subjects,17 had oral exams at entry but not week 2: 11 premature discontinuation, 2 missed visits, and 4 without specific reasons. 204 subjects received oral exams at both entry and week 2. 2 more participants were excluded from the final analysis because they had no pseudomem candi at entry, which led to a total of 202 subjects.
Measure: Number; unit: participants
Arm/Group | Arm A: Topical GV Solution | Arm B: Nystatin Oral Suspension
Number analyzed (Participants) | 100 | 102
participants | 76 | 73
Statistical Analysis 1: Comparison: Arm A: Topical GV Solution vs Arm B: Nystatin Oral Suspension; Repeated confidence intervals (RCIs) were used to control type I error.A interim analysis was conducted by a 99.7% CI. The final analyses use a 95.1% CI, based on the Lan-DeMets error-spending function corresponding to the O'Brien-Fleming boundary.76% of 100 participant in arm GV had cure or improvement of OC after 14 days of treatment, and 71.6% of 102 in arm nystatin had cure or improvement of OC. Difference in clinical efficacy rates between GV and nystatin 95.1% CI is 0.044 (-0.077, 0.166); Test type: Superiority or Other; Difference in proportion with clinical e = 0.044, 95.1% CI 2-sided [-0.077 to 0.166]

2. Secondary Outcome: Number of Participant With Symptom
Description: Symptoms were assessed using a visual analog scale where the level of discomfort and pain were recorded and quantified using a scoring system from 0 to 3. 0=no discomfort/pain; 1=mild discomfort/pain; 2=Moderate discomfort/pain; 3=Severe discomfort/pain.
Time Frame: after 14 days of treatment
Population: At entry, a total of 217 observations (106 in GV arm; 111 in nystatin arm) were available to evaluate the symptoms (pain and discomfort) associated with OC. At the end of treatment, a total of 204 observations were available to evaluate the symptoms associated with OC using extended Mantel-Haenszel test between GV and nystatin arms.
Measure: Number; unit: participants
Arm/Group | Arm A: Topical GV Solution | Arm B: Nystatin Oral Suspension
Number analyzed (Participants) | 106 | 111
participants
  Pain at entry | 106 | 111
  Pain at end of treatment | 102 | 102
  Discomfort at entry | 106 | 111
  Discomfort at end of treatment | 102 | 102

3. Secondary Outcome: Quantitative Yeast Colony Counts
Description: If quantitative yeast culture yielding < 20 CFU/mL of Candida spp., then we call this mycological success
Time Frame: At weeks 0, 2, 6
Population: At entry, 210 observations were available (182 had positive culture result for Candida specimen, and 175 of those had colony count performed) to evaluate quantitative yeast colony counts.
  N= 78 (GV), 70 (Nystatin) at end of treatment; N= 51 (GV), 35 (Nystatin) at week 6;
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Arm A: Topical GV Solution | Arm B: Nystatin Oral Suspension
Number analyzed (Participants) | 88 | 87
CFU/mL
  At entry, week 0 | 7.2497 (2.2382) | 7.0037 (2.0584)
  At end of treatment (week 2) | 6.9374 (2.1438) | 5.8888 (2.3970)
  At week 6 | 6.7388 (2.3469) | 6.5929 (2.3668)

4. Secondary Outcome: Tolerance
Description: The investigators will measure tolerance using a scale from 0 to 3 (0=No side effects experienced, no changes in treatment; 1=Some side effects experienced, but not enough to modify treatment; 2=Some side effects experienced, resulted in treatment interruption; 3=Side effects experienced, resulted in treatment discontinuation.)
Time Frame: After 14 days of treatment
Population: The analysis for tolerance was based on 208 observations.
Measure: Number; unit: participants
Arm/Group | Arm A: Topical GV Solution | Arm B: Nystatin Oral Suspension
Number analyzed (Participants) | 103 | 105
participants
  No side effects, no changes in treatment | 100 | 98
  Some side effects, no changes in treatment | 3 | 6
  Some side effects, treatment interruption | 0 | 1

5. Secondary Outcome: Number of Participants Who Were Adherent.
Description: Adherence was reported as a dichotomous variable (adherence vs. non-adherence). Participants who have missing doses less than 15% will be considered as adherent, i.e., if a participant is in the GV arm, then the cutoff point is 28*0.15=4 doses; and for the nystatin arm is 56*0.15=8 doses.
Time Frame: After 14 days of treatment
Population: The analysis for adherence was based on 209 observations.
Measure: Number; unit: participants
Arm/Group | Arm A: Topical GV Solution | Arm B: Nystatin Oral Suspension
Number analyzed (Participants) | 104 | 105
participants
  Adherent | 95 | 95
  Non-adherent | 9 | 10

6. Secondary Outcome: Self-Assessment of General Health
Description: Participants rated their general health on two scales. One is a five point scale ranging from 1 to 5 (1=Excellent; 2=Very Good; 3=Good; 4=Fair; 5=Poor)
Time Frame: Weeks 0, 6
Population: N=110 (GV), 110 (Nystatin) wk 0 N= 96 (GV), 95 (Nystatin) wk 6
Measure: Number; unit: participants
Arm/Group | Arm A: Topical GV Solution | Arm B: Nystatin Oral Suspension
Number analyzed (Participants) | 110 | 110
participants
  Week 0: Excellent | 1 | 4
  Week 0: Very Good | 13 | 11
  Week 0: Good | 52 | 56
  Week 0: Fair | 39 | 30
  Week 0: Poor | 5 | 9
  Week 6: Excellent | 5 | 7
  Week 6: Very Good | 29 | 25
  Week 6: Good | 42 | 42
  Week 6: Fair | 18 | 18
  Week 6: Poor | 2 | 3

7. Secondary Outcome: Number of Participants Who Found GV and Nystatin Acceptable.
Description: Acceptability was defined as the willingness to use the drug if it is proven effective to treat oral candidiasis. Participants were asked whether or not they would be willing to use the assigned treatment via questionnaires.
Time Frame: After 14 days of treatment
Population: The analysis for acceptability of treatment was based on 209 subjects.
Measure: Number; unit: participants
Arm/Group | Arm A: Topical GV Solution | Arm B: Nystatin Oral Suspension
Number analyzed (Participants) | 104 | 105
participants | 100 | 98

ADVERSE EVENTS:
Time Frame: From entry (week 0) to end of study.
Description: The protocol requested reporting of grade 3 or higher of adverse events and any adverse event that led to a change in study treatment, regardless of grade. Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009), was used for grading
Groups:
- Gentian Violet: Topical GV 0.00165% solution (5 mL swish and gargle for 1 minute and expectorate [spit] 2 times per day [BID]) for 14 days
  Gentian Violet: Participants will be administered topical Gentian violet solution, orally, twice daily for 14 days.
- Nystatin: Nystatin oral suspension (5 mL of 100,000 units/mL swish for 1 minute and swallow 4 times per day [QID]) for 14 days
  Nystatin oral suspension: Participants will be administered Nystatin oral suspension 4 times a day for 14 days.
Arm/Group | Gentian Violet | Nystatin
Serious Adverse Events (participants affected / at risk) | 18/110 | 17/111
Other Adverse Events (participants affected / at risk) | 103/110 | 101/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gentian Violet (N=110) | Nystatin (N=111)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Death (General disorders) | 2 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Encephalitis viral (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1
HIV infection WHO clinical stage IV (Infections and infestations) | 1 | 0
Malaria (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 2
Meningitis cryptococcal (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 3 | 2
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Nephropathy (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gentian Violet (N=110) | Nystatin (N=111)
Cheilitis (Gastrointestinal disorders) | 9 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 6
Leukoplakia oral (Gastrointestinal disorders) | 6 | 4
Odynophagia (Gastrointestinal disorders) | 6 | 3
Oral disorder (Gastrointestinal disorders) | 11 | 14
Oral mucosal erythema (Gastrointestinal disorders) | 5 | 8
Stomatitis (Gastrointestinal disorders) | 7 | 6
Chest pain (General disorders) | 8 | 10
Pyrexia (General disorders) | 5 | 9
Oral candidiasis (Infections and infestations) | 31 | 26
Oral hairy leukoplakia (Infections and infestations) | 6 | 11
Pneumonia bacterial (Infections and infestations) | 5 | 8
Pulmonary tuberculosis (Infections and infestations) | 9 | 6
Alanine aminotransferase increased (Investigations) | 12 | 6
Aspartate aminotransferase increased (Investigations) | 31 | 26
Blood albumin decreased (Investigations) | 58 | 53
Blood alkaline phosphatase increased (Investigations) | 18 | 11
Blood bicarbonate decreased (Investigations) | 21 | 20
Blood calcium decreased (Investigations) | 43 | 50
Blood creatinine increased (Investigations) | 7 | 5
Blood glucose decreased (Investigations) | 1 | 6
Blood glucose increased (Investigations) | 7 | 9
Blood magnesium decreased (Investigations) | 11 | 10
Blood phosphorus decreased (Investigations) | 10 | 10
Blood potassium decreased (Investigations) | 9 | 11
Blood sodium decreased (Investigations) | 52 | 37
Blood uric acid increased (Investigations) | 10 | 20
Haemoglobin decreased (Investigations) | 33 | 33
Neutrophil count decreased (Investigations) | 22 | 29
White blood cell count decreased (Investigations) | 17 | 23
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No